CLINICAL TRIAL: NCT00451581
Title: A Prospective Randomized Multicenter Study Comparing Different Dilation Durations During Endoscopic Papillary Balloon Dilatation for Bile Duct Stones.
Brief Title: A Prospective Randomized Study Comparing Different Dilation Durations for Endoscopic Papillary Balloon Dilatation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9561709036
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2006-10

CONDITIONS: Choledocholithiasis
Keywords: Endoscopic papillary balloon dilatation; Endoscopic sphincterotomy; Choledocholithiasis; Efficacy; Complication
MeSH Terms: conditions — Choledocholithiasis

INTERVENTIONS:
Procedure: Endoscopic papillary balloon dilation-5 minutes
Procedure: Endoscopic papillary balloon dilation-1 minute

SUMMARY:
Endoscopic papillary balloon dilation is as effective as sphincterotomy in treating bile duct stone. However, a need to switch to sphincterotomy is noted in about 20% of cases receiving dilation for lithotripsy. It is hypothesized that a longer dilation duration (5 min. vs. 1 min.) can decrease the need of switching to sphincterotomy.

DETAILED DESCRIPTION:
Endoscopic papillary balloon dilatation (EPBD) has been proposed as an alternative to endoscopic sphincterotomy (EST) for endoscopic treatment of common bile duct (CBD) stones. EPBD is as effective as EST in stone clearance with a lower risk of hemorrhage, and may preserve the function of sphincter of Oddi. However, it has been reported that about 20% of patients undergoing EPBD need EST as a rescue procedure for lithotripsy. A longer dilation duraton of 5 mintues as opposed to 1 minute has been proposed to decrease oozing after dilation and facilitate lithotripsy, and it is hypothesized that it will reduce the need of switching to EST.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endoscopic retrograde cholangiopancreatography for choledocholithiasis

Exclusion Criteria:

* Consent not obtained.
* No apparent stone.
* Intradiverticular papilla.
* Prior EST.
* Bile duct stricture.
* Pancreatic or biliary malignant disorders.
* Intrahepatic stones.
* Active acute pancreatitis.
* Sphincter of Oddi dysfunction.
* Pregnancy.
* Primary sclerosing cholangitis or choledochocyst.
* Previous biliary surgery other than cholecystectomy.
* Stone impaction at ampulla.
* Precut for cannulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2007-01; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
need of switching to sphincterotomy

SECONDARY OUTCOMES:
efficacy of lithotripsy
post-ERCP complications

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chih Liao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] 1. Bergman JJ, Rauws EA, Fockens P, van Berkel AM, Bossuyt PM, Tijssen JG, Tytgat GN, Huibregtse K. Randomised trial of endoscopic balloon dilation versus endoscopic sphincterotomy for removal of bileduct stones. Lancet 1997;349:1124-9. 2. Komatsu Y, Kawabe T, Toda N, Ohashi M, Isayama M, Tateishi K, Sato S, Koike Y, Yamagata M, Tada M, Shiratori Y, Yamada H, Ihori M, Kawase T, Omata M. Endoscopic papillary balloon dilation for the management of common bile duct stones: experience of 226 cases. Endoscopy 1998;30:12-7. 3. Lin CK, Lai KH, Chan HH, Tsai WL, Wang EM, Wei MC, Fu MT, Lo CC, Hsu PI, Lo GH. Endoscopic balloon dilatation is a safe method in the management of common bile duct stones. Dig Liver Dis 2004;36:68-72.
- [Derived] Liao WC, Lee CT, Chang CY, Leung JW, Chen JH, Tsai MC, Lin JT, Wu MS, Wang HP. Randomized trial of 1-minute versus 5-minute endoscopic balloon dilation for extraction of bile duct stones. Gastrointest Endosc. 2010 Dec;72(6):1154-62. doi: 10.1016/j.gie.2010.07.009. Epub 2010 Sep 25. PMID 20869710